CLINICAL TRIAL: NCT06687148
Title: Global Changes Associated With Sacroiliac Joint Dysfunction and Its Reversal by Manipulation - Pilot Study
Brief Title: Global Changes Associated With Sacroiliac Joint Dysfunction
Acronym: GCASID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Luís Filipe Albuquerque, Principal Investigator, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Global changes with SIJD
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Sacroiliac Dysfunction
Keywords: manipulative intervention; pain; muscle tone; semiology of sacroiliac dysfunction
MeSH Terms: conditions — Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Manipulative therapy (Experimental): Experimental group, subject to manipulation performed by the same Physiotherapist, using the techniques described by Shadmehr, A. et al (2018).
  Interventions: Other: Manual manipulation
- Participants will be submitted to a simulated manipulation. (Sham Comparator): Sham group, subjected only to a simulation of manipulation, using the same gestures, but without manipulating, used as a placebo group.
  Interventions: Other: Sham manipulation
- Group will not be subject to any intervention. (No Intervention): Control group, which will not be subject to any intervention.

INTERVENTIONS:
Other: Manual manipulation — The participants will receive one session of manipulation if in the experimental group. It should be mentioned that the technique will be carried out by a physiotherapist with a history of more than 10 years of manual therapy. For instance, to correct right anterior innominate rotation, the participant will be made to lie on the side so that the affected side is upward. The physiotherapist will stand in front of the participant; first we will put their shoulders, pelvis and lower limbs in neutral position and place the right hand on the anterior superior iliac spine (ASIS) and the left hand on the ischium tuberosity and with a rotational movement of the hands, the physiotherapist will rotate the ilium posteriorly. At the end of the range, we will replace the position of hands and place the left forearm on the ischium tuberosity and place the right hand on the upper participant's shoulder and will move it toward the bed at the end of the range in exhalation a thrust will be executed.
  Arms: Manipulative therapy
Other: Sham manipulation — The participants will receive one session of sham manipulation if in the sham group. For instance, to correct right anterior innominate rotation, the participant will be made to lie on the side so that the affected side is upward. The physiotherapist will stand in front of the participant; first we will put their shoulders, pelvis and lower limbs in neutral position and place the right hand on the anterior superior iliac spine (ASIS) and the left hand on the ischium tuberosity and with a rotational movement of the hands, the physiotherapist will rotate the ilium posteriorly. At the end of the range, we will replace the position of hands and place the left forearm on the ischium tuberosity and place the right hand on the upper participant's shoulder and will move it toward the bed at the end of the range in exhalation, the physiotherapist will pretend to execute a thrust.
  Arms: Participants will be submitted to a simulated manipulation.

SUMMARY:
* Summary Sacroiliac joint dysfunction (ASI) is an alteration in the normal biomechanics of the joint, which leads to hypomobility or hypermobility of that joint. It is one of the most common causes of misdiagnosis in low back pain and when not treated correctly, it often evolves into chronic pain (30% to 42%) and disability. Manipulating the dysfunctional ASI appears to result in benefits and significantly positive changes at various levels, in all segments of the human body. With this investigation, we intend to clarify and deepen the possible correlation between the changes that normally accompany this dysfunction, as well as its possible reversibility with its normalization.
* Objectives

The investigators will essentially have two main objectives:

1. Mapping of the most evident symptomatic changes, when sacroiliac joint dysfunction is present, in terms of pain and muscle tone;
2. To try to understand the immediate, global and immediate effect of ASI manipulation.

   * Study design Quantitative, with experimental study design, with the sample comprising individuals with SIJ dysfunction, where all participants will be randomly allocated to the experimental, control and sham groups. It will be carried out at the University of Aveiro facilities.

Initially, we will assess the participants with sacroiliac dysfunction. The experimental will be manipulated, the control group will do nothing, and the sham group will be submitted to a hypothetical manipulation (sham manipulation). Consequently, the patients will be assessed again, measuring the subjective and objective degree of pain and muscle tone.

- Material and methods

We will make use of:

* Standing flexion test;
* Sitting Flexion Test;
* Faber Test;
* EVA , to subjectively assess pain;
* Pressure algometer, to objectively assess pain ;
* MyotonPro, to assess muscle tone;

DETAILED DESCRIPTION:
Introduction

ASI dysfunction refers to a state of altered biomechanics of this joint . This dysfunction can result from repetitive stress , degeneration, lumbar deformities, inflammation, and previous lumbar fusion.

ASI dysfunction is an alteration in the normal biomechanics of the joint, which leads to hypomobility or hypermobility of that joint. It is one of the most common causes of misdiagnosis in low back pain and when not treated correctly, it often develops into chronic pain (30% to 42%) and disability.

The SIJ has a crucial function in mobility, stability and resistance against shear forces, and is also wrongly undervalued as the origin of low back pain and, with the increase in average life expectancy, it has become an extremely prevalent problem.

Manipulation of the SIJ in dysfunction appears to bring about benefits and significantly positive changes at various levels. The analysis of the results of two manipulative therapy techniques in patients with sacroiliac dysfunction revealed a statistically significant improvement immediately after treatment, after 48 hours and one month later, in terms of both pain and disability, as favourable developments were recorded in measurements using the VAS and the Oswestry Disability Index (ODI).

Even in asymptomatic individuals, there seem to be changes that are not just local, when manipulating the ASI, they came to the conclusion that the manipulation of the ASI applied bilaterally in asymptomatic people resulted in immediate changes in load distribution on the plantar support, in the orthostatic position, after baropodometric analysis using a force platform.

The benefits of this therapeutic approach were also defended, after a study in young females with SIJ dysfunction, subjected to a single SIJ manipulation session, in which the analysis of results after evaluation with EVA instruments and a digital algometer ( Model J- Tech ), indicate that the manipulation helped to alleviate the level of pain, with the effects lasting for 24 hours, immediately increasing the range of motion of internal and external rotations of the hips and lumbar flexion and extension.

Despite the existence of multiple studies on the benefits of this type of approach at various levels, in a more or less localized way, we did not find any study that showed correlated changes at a global level. With this work, we will seek to map the most evident symptomatological changes in the different regions of the human body associated with ASI dysfunction and evaluate the potential of manipulating the ASI in individuals with dysfunction of this joint, analyzing at specific points in the different segments, the initial state in terms of inequality of perceived pain and difference in muscle tone verified, measuring, following manipulation, the observable changes in these variables. As instruments for this assessment, we will use the following variables:

1. Pain - EVA and Pressure Algometer;
2. Muscle tone - MyotonPro ;

The main objective of this PhD thesis will be to understand the effect of manipulation on the dysfunction of the SIJD.

Objectives

1. Mapping of the most evident symptomatological changes, when sacroiliac joint dysfunction is present, in terms of pain and muscle tone;
2. To study the immediate effect of ASI manipulation and the hypothetical correlation with the changes recorded, in pain level and muscle tone.

Study Design and Methods

Study Design Experimental pilot study, where participants will be randomly allocated to experimental, control and sham groups. It will be carried out at the University of Aveiro facilities, with a sample of 21 students.

Participants The study sample will be a convenience sample, randomly selected from the universe of students at the University of Aveiro, invited to participate in the study.

* Inclusion criteria: young adults, of both sexes, aged between 18 and 30 years, with sacroiliac joint dysfunction demonstrated by standing flexion test, sitting flexion test and strength test with applied kinesiology.
* Exclusion criteria: students of the Bachelor's Degree in Physiotherapy, Individuals with neurological injuries, under the effect of local anesthetics, or subject to another type of therapeutic intervention, during the intervention period.
* Ethical considerations: All volunteers will be informed about the objectives of the study, procedures, methods of data collection and processing/confidentiality, as well as the possible benefits and harms. They will have the possibility to refuse participation at any time, and will be required to express their consent in light of the protocol of the Declaration of Helsinki.

Variables :

* Pain (EVA and algometer);
* Muscle tone (Myoton Pro).

Instruments : -

* EVA , to assess the subjective sensation of pain perceived by the participant;
* Pressure Algometer , to assess pain, used at the following points:

  * Lower limbs: muscular belly of the external calves, 8 cm below their origin and muscular belly of the internal calves, 12 cm below the insertion, cuboids and tarsal naviculars;
  * Upper limbs: bilaterally at the level of the muscular belly of the short portion of the biceps brachii, 9 cm above the elbow crease and muscular belly of the brachialis, 3 cm below the vertex of the V deltoid;
  * Cervical spine: At the level of the transverse processes of C4, bilaterally;
  * Lumbar spine: At the level of the transverse processes of L3, bilaterally;
  * Sacroiliac joints bilaterally, at the level of the posterior superior iliac spine, bilaterally;
  * Craniocervical transition, bilaterally, at the level of the occipital origin of the upper trapezius muscle;
  * External and internal joint interline, middle third, in both knees;
  * Iliac fossa bilaterally, 5 cm internally to the anterior superior iliac spine;
  * Transition from the hypochondrium to the lateral abdominal region, bilaterally;
* MyotonPro : at the same points used with the pressure algometer, at the level of the upper and lower limbs, to assess muscle tone.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of sacroiliac joint dysfunction.

Exclusion Criteria:

* Students of the Bachelor's Degree in Physiotherapy;
* Individuals with neurological injuries:
* Under the effect of local anesthetics;
* Subject to another type of therapeutic intervention, during the intervention period.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Pain | From enrollment the assessment will be executed, before and immediately after the intervention taking approximately one week
  Pain will be assessed with the Visual Analogue Scale (VAS), with a horizontal line graded 0 (no pain) to 10 (worse pain).
Myotonometric assessment of muscular tonus | From enrollment the assessment will be executed, before and immediately after the intervention taking approximately one week
  The investigators measure the muscle tone with the device Myoton Pro
Pain assessment with algometry | From enrollment the assessment will be executed, before and immediately after the intervention taking approximately one week
  Pressure algometer

CONTACTS AND LOCATIONS:
Locations (1):
- Aveiro University, Aveiro, Aveiro District, Portugal

REFERENCES:
- [Background] Kamali F, Shokri E. The effect of two manipulative therapy techniques and their outcome in patients with sacroiliac joint syndrome. J Bodyw Mov Ther. 2012 Jan;16(1):29-35. doi: 10.1016/j.jbmt.2011.02.002. Epub 2011 Mar 11. PMID 22196424
- [Background] Grieve E. Lumbo-pelvic rhythm and mechanical dysfunction of the sacro-iliac joint. Physiotherapy. 1981 Jun;67(6):171-3. No abstract available. PMID 7301975
- [Background] Gartenberg A, Nessim A, Cho W. Sacroiliac joint dysfunction: pathophysiology, diagnosis, and treatment. Eur Spine J. 2021 Oct;30(10):2936-2943. doi: 10.1007/s00586-021-06927-9. Epub 2021 Jul 16. PMID 34272605